CLINICAL TRIAL: NCT03918603
Title: Reduction of Mechanical Ventilation-induced Lesions During ARDS With Multimodal Ultra-protective Ventilation in Combination With ECMO
Brief Title: Decrease of Lesions Induced by Mechanical Ventilation During ARDS
Acronym: ECMO-VILI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: mid-term analysis
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-45; 2018-A02297-48 (Registry Identifier: APHM)
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra-protective multimodal ventilation group (Experimental): Patient will be diposed on ventral decubitus: one session at least more than 12 hours between inclusion and H48
  Interventions: Other: ventral décubitus
- protective ventilation group (No Intervention): Patient will received usual care

INTERVENTIONS:
Other: ventral décubitus — Patient will have one session at least more than 12 hours between inclusion and H48 of ventral décubitus
  Arms: ultra-protective multimodal ventilation group

SUMMARY:
Modification of mechanically ventilated lesions by an ultra-protective multimodal strategy compared to a protective strategy in patients with veno-venous ECMO for severe ARDS.

DETAILED DESCRIPTION:
the hypothesis is that ECMO, in addition to improving gas exchange, should limit the deleterious effects of mechanical ventilation (mechanical ventilation-induced lesions, VILI) by drastically reducing minute ventilation (volume reduction). current, Vt, reduction of respiratory rate, reduction of mechanical power, reduction of motor pressure or driving pressure), adapting the level of PEEP from the data collected by monitoring oesophageal pressure and systematically performing positioning sessions in the prone position. This ultra-protective strategy could thus promote the restoration of the integrity of the alveolo-capillary membrane and thus facilitate the healing of patients. In order to verify this concept and, if necessary, to propose a study whose objectives would be more clinical (mortality, ventilator-free days), we propose to carry out a study aimed at showing that this ultra-protective multimodal strategy reduces the lesions induced by mechanical ventilation compared to usual protective ventilatory management during the ECMO as proposed in the EOLIA study.

ELIGIBILITY:
Inclusion Criteria:

* severe ARDS with a PaO2 / FiO2 ratio ≤ 70 mmHg (for at least 2h) measured at PEEP> 10 cmH2O and FiO2 = 1
* OR a severe ARDS with a PaO2 / FiO2> 70 ratio but <100 mmHg with a plateau pressure> 35 cmH2O and a pH <7.20

Exclusion Criteria:

* Patients with associated hemodynamic failure requiring veno-arterial ECMO
* Impossibility of setting up or contraindication to the placement of an esophageal tube
* Impossibility of realization of ventral decubitus
* Patient to receive corticosteroids during the first 48 hours following venous venous ECMO.
* Patients assisted by veno-venous ECMO for more than 24 hours.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
inflammation of biotrauma | 36months
  Interleukine dosage in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Guervilly C, Fournier T, Chommeloux J, Arnaud L, Pinglis C, Baumstarck K, Boucekine M, Valera S, Sanz C, Adda M, Bobot M, Daviet F, Gragueb-Chatti I, Forel JM, Roch A, Hraiech S, Dignat-George F, Schmidt M, Lacroix R, Papazian L. Ultra-lung-protective ventilation and biotrauma in severe ARDS patients on veno-venous extracorporeal membrane oxygenation: a randomized controlled study. Crit Care. 2022 Dec 12;26(1):383. doi: 10.1186/s13054-022-04272-x. PMID 36510324